CLINICAL TRIAL: NCT06974786
Title: Frontline T-cell Engager vs Autologous Stem Cell Transplant and Measurable Residual Disease (MRD)-Guided Sequential Intensification thERapy in Multiple Myeloma (FASTER)
Brief Title: Frontline T-cell Engager vs Autologous Stem Cell Transplant (ASCT) and Measurable Residual Disease (MRD)-Guided Sequential Intensification thERapy in Multiple Myeloma
Acronym: FASTER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Pfizer (Industry); coMMit, Myeloma Trials, Innovated (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MM 195
Record Dates: First submitted 2025-05-06; First posted 2025-05-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma, Newly Diagnosed; Multiple Myeloma (MM)
Keywords: MM; Newly diagnosed multiple myeloma; NDMM; MRD; ASCT; T-cell engager; Elranatamab; Daratumumab; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A (Elranatamab + Daratumumab) (Experimental): Participants will receive step up dosing of Elranatamab subcutaneously in first cycle followed by weekly dosing for the remainder of the cycle 1. In cycle 2 and 3, elranatamab will be administered every two weeks (Consolidation portion). This will be followed by elranatamab every 4 weeks for 12 cycles in the Maintenance 1 portion. Daratumumab will be given subcutaneously at a fixed dose every 4 weeks starting at Cycle 2 and 3 of Consolidation and for 12 cycles in the Maintenance 1 portion of the study. After completion of Maintenance 1, participants with MRD negativity will receive Elranatamab monotherapy every 4 weeks for additional 12 cycles in Maintenance 2 portion. Participants with MRD positivity will proceed to Arm A1. Participants will undergo therapy in the assigned arm until disease progression, permanent discontinuation (irrespective of reason), death or completion of planned therapy. Cycles will be 28 days. Consolidation consists of 3 cycles; Maintenance 1 consists of 12
  Interventions: Drug: Elranatamab; Drug: Daratumumab
- Arm B (ASCT + lenalidomide/daratumumab) (Active Comparator): Participants will undergo ASCT according to standard of care institutional practices in the Consolidation portion of the study followed by twelve 28-day cycles of Lenalidomide and Daratumumab in the Maintenance 1 portion. After completion of Maintenance 1, participants with MRD negativity will receive Lenalidomide monotherapy for additional 12 cycles in Maintenance 2 portion. Participants with MRD positivity will proceed to Arm B1. Participants will undergo therapy in the assigned arm until disease progression, permanent discontinuation (irrespective of reason), death or completion of planned therapy. Cycles will be 28 days. Consolidation consists of ASCT; Maintenance 1 consists of 12 cycles; Maintenance 2 consists of 12 cycles. Up to 50 participants will be enrolled to this arm.
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Procedure: autologous stem cell transplantation
- Arm A1 (Late Intensification) (Experimental): Participants randomized to Arm A that have MRD positivity after Maintenance 1 will undergo ASCT according to standard of care institutional practices followed by twelve 28-day cycles of maintenance treatment with Lenalidomide and Daratumumab in the Late Intensification portion of the study.
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Procedure: autologous stem cell transplantation
- Arm B1 (Late Intensification) (Experimental): Participants randomized to Arm B that have MRD positivity after Maintenance 1 will receive Elranatamab in combination with Daratumumab for three 28-day cycles as consolidation, followed by Elranatamab in combination with Daratumumab for additional twelve 28-day cycles of maintenance treatment in the Late Intensification portion of the study.
  Interventions: Drug: Elranatamab; Drug: Daratumumab

INTERVENTIONS:
Drug: Elranatamab — Participants will receive step up dosing of Elranatamab subcutaneously in first cycle of consolidation followed by fixed dosing for 2 additional cycles and for 12 cycles in maintenance. Arm A participants will receive additional 12 cycles of Elranatamab monotherapy if they are MRD negative after Maintenance 1 for a total of 27 cycles. Cycles will be 28 days.
  Other Names: Elrexfio
  Arms: Arm A (Elranatamab + Daratumumab); Arm B1 (Late Intensification)
Drug: Daratumumab — Participants will be given 1800 mg of Daratumumab subcutaneously every 4 weeks for up a maximum of 26 cycles.
  Other Names: Darzalex
Drug: Lenalidomide — Participants will receive 10 mg of Lenalidomide daily by mouth for 21 days of each 28-day cycle for up to a maximum of 24 cycles.
  Other Names: Revlimid
  Arms: Arm A1 (Late Intensification); Arm B (ASCT + lenalidomide/daratumumab)
Procedure: autologous stem cell transplantation — Participants will undergo ASCT as standard treatment following individual site's processes and practices.
  Other Names: ASCT
  Arms: Arm A1 (Late Intensification); Arm B (ASCT + lenalidomide/daratumumab)

SUMMARY:
This is an open-label, multi-site, Phase II randomized trial with response-adaptive design for newly diagnosed multiple myeloma (NDMM) participants who have had prior induction therapy. The primary objective of this study is to compare the rates of achieving undetectable measurable residual disease (MRD) in the bone marrow with elranatamab and daratumumab employed as post-induction consolidation and maintenance treatment (Arm A) versus autologous stem cell transplant (ASCT) followed by lenalidomide and daratumumab treatment (Arm B).

DETAILED DESCRIPTION:
This is an open-label, multi-site, Phase II randomized trial with response-adaptive design for newly diagnosed multiple myeloma (NDMM) participants who had prior induction therapy with one proteasome inhibitor, lenalidomide, and an anti-CD38 Monoclonal antibody (mAb) for 16-24 weeks and obtained at least partial response (PR). Eligible participants will be randomized in equal allocation to receive either elranatamab and daratumumab as consolidation and maintenance treatment (Arm A) or to undergo autologous stem cell transplant (ASCT) followed by lenalidomide and daratumumab maintenance treatment (Arm B). Patients who have residual detectable disease by MRD assessment after one year of consolidation and maintenance will undergo "late intensification" and receive the alternative therapy. Patients who achieve sustained "MRD-negativity" on 2 consecutive assessments will discontinue treatment with observation for disease progression or MRD resurgence. Elranatamab is a humanized bispecific antibody which binds to BCMA on MM cells and CD3 on T cells. Elranatamab activates and directs T cells to induce a cytotoxic T-cell response against myeloma cells. Daratumumab is a CD-38 directed therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years with no upper age limit.
2. Newly diagnosed multiple myeloma with indication for initiation of therapy diagnosed within last 12 months. Pretreatment parameters necessary for disease characterization and response assessment must be available.
3. Eligible for ASCT according to institutional policy as evaluated by investigator.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Appendix A).
5. Prior induction therapy including one PI, lenalidomide, and an anti-CD38 mAb for 16-24 weeks, obtaining at least a partial response (PR).
6. Measurable disease meeting at least 1 of the following criteria (at the time of diagnosis):

   a. Serum monoclonal (M) protein ≥1.0 g/dl (≥0.5 g/dl if IgA, IgD, IgE or IgM MM).

   b. ≥200 mg of M protein/24h in the urine. c. Difference between affected and unaffected free light chain ≥10 mg/dL with abnormal kappa to lambda ratio.
7. Have trackable clonogenic sequence using ClonoSEQ® (Seattle, WA) identified from a high disease burden sample obtained as SoC and enabling MRD testing during screening phase.
8. Have clinical laboratory values meeting the following criteria during the Screening Phase and also at start of administration of study treatment:

   • Hemoglobin ≥8g/dL without prior red blood cells (RBC) transfusion within 14 days before the laboratory test; recombinant human erythropoietin use is permitted

   • Platelets ≥75,000/µl

   • Absolute neutrophil count ≥1,000/µl (prior growth factor support is permitted but must be without support for 7 days for granulocyte colony stimulating factor (G-CSF) or granulocyte-macrophage colony stimulating Factor (GM-CSF) and for 14 days for pegylated G-CSF before screening lab test

   • Aspartate aminotransferase and alanine aminotransferase ≤2.5 × upper limit of normal (ULN)
   * Renal function: Creatinine clearance (CrCl) ≥40 mL/min based on calculation using Cockcroft-Gault formula or measured by a 24-hour urine collection.
   * Total bilirubin ≤2 × ULN, except in participants with congenital bilirubinemia, such as Gilbert syndrome (in which case direct bilirubin ≤3 × ULN is required)
   * Serum calcium corrected for albumin ≤14 mg/dL (≤3.5 mmol/L) or free ionized calcium ≤6.5 mg/dL (≤1.6 mmol/L)
9. Achievement of at least PR to induction therapy, without prior progression of disease.
10. Prior completion of standard of care mobilization and collection of stem cells (minimum 2 × 106 CD34+ cells/kg) without use of chemotherapy mobilization, any time prior to or during screening phase.
11. A woman of childbearing potential must have a negative highly sensitive serum pregnancy test at screening and again within 24 hours of the start of study treatment and must agree to further serum or urine pregnancy tests during the study.
12. A woman must be:

    a. Not of childbearing potential, or b. Of childbearing potential and practicing true abstinence; or i. Have a sole partner who is vasectomized; or ii. Practicing ≥1 highly-effective, user-independent method of contraception (Appendix B) NOTE: Participant must agree to continue the above throughout the study and for 4 months after the last dose of study treatment. If a woman becomes of childbearing potential after start of the study the woman must comply with point (b) as described above.
13. A woman must agree not to donate eggs (ova, oocytes) or freeze for future use, for the purposes of assisted reproduction during the study and for 4 months after receiving the last dose of study treatment.
14. A man must wear a condom (with or without spermicidal foam/gel/film/cream/suppository) when engaging in any activity that allows for passage of ejaculate to another person during the study and for a minimum of 90 days after receiving the last dose of study treatment. If a female partner is of childbearing potential, she must also be practicing a highly effective method of contraception.

    NOTE: If the male participant is vasectomized, he still must wear a condom (with or without spermicidal foam/gel/film/cream/suppository), but his female partner is not required to use contraception.
15. A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 90 days after receiving the last dose of study treatment.
16. Must be willing and able to adhere to the lifestyle restrictions specified in this protocol.
17. Must sign an Informed Consent Form (ICF) (or their legally acceptable representative must sign) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study.
18. All participants must agree to comply with and be enrolled in Revlimid Risk Evaluation and Mitigation Strategy (REMS) program.
19. All participants must agree to comply with and be enrolled in elranatamab Risk Evaluation and Mitigation Strategy (REMS) program.
20. All participants must meet institution-specific criteria for ASCT eligibility as assessed by the Investigator.

Exclusion Criteria:

1. Diagnosis of primary light chain amyloidosis, POEMS, Waldenstrom's macroglobulinemia, plasma cell leukemia, or central nervous system (CNS) involvement by MM.
2. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients (refer to the elranatamab Investigator's Brochure [IB] and appropriate package inserts).
3. Prior or concurrent exposure to any of the following:

   c. Any anti-BCMA therapy. d. Epigenetic therapy, or treatment with an investigational drug or an invasive investigational medical device within 21 days or ≥5 half-lives, whichever is less.

   e. Investigational vaccine within 4 weeks. f. Live, attenuated vaccine within 4 weeks before randomization. g. Radiotherapy within 14 days. h. Gene-modified adoptive cell therapy (e.g., CAR modified T cells, NK cells). i. Cytotoxic therapy within 14 days.
4. Minimum washout period for prior therapy:

   1. PI therapy - 14 days.
   2. IMiD agent therapy -14 days.
   3. Anti CD38 monoclonal therapy - 14 days.
   4. Corticosteroids - 7 days.
5. Known active CNS involvement or exhibits clinical signs of meningeal involvement of MM. If either is suspected, negative whole brain magnetic resonance imaging and lumbar cytology are required.
6. Myelodysplastic syndrome or active malignancies (i.e., progressing or requiring treatment change in the last 24 months) other than MM. The only allowed exceptions are:

   a. Non-muscle invasive bladder cancer treated within the last 24 months that is considered completely cured.

   b. Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured.

   c. Non-invasive cervical cancer treated within the last 24 months that is considered completely cured.

   d. Localized prostate cancer (N0M0): i. With a Gleason score of ≤6, treated within the last 24 months, or untreated and under surveillance.

1) With a Gleason score of 3+4 that has been treated >6 months prior to full study screening and considered to have a very low risk of recurrence, or e. History of localized prostate cancer and receiving androgen deprivation therapy and considered to have a very low risk of recurrence.

f. Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer and receiving antihormonal agents and considered to have a very low risk of recurrence (<5% over 5 years).

g. Other malignancy that is considered cured with minimal risk of recurrence. 7. Stroke or seizure within 6 months prior to signing ICF. 8. Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 is <50% of predicted normal.

9. Moderate or severe persistent asthma within the past 2 years or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.

10. Prior allogeneic bone marrow, hematopoietic stem cell or solid organ transplant.

11. Participant is pregnant, breast-feeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of study treatment.

12. Participant plans to father a child while enrolled in this study or within 90 days after the last dose of study treatment.

13. Presence of the following cardiac conditions: h. New York Heart Association Class III or IV congestive heart failure i. Myocardial infarction or coronary artery bypass graft ≤6 months prior to randomization j. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration.

k. History of severe non-ischemic cardiomyopathy. 14. Any of the following:

1. History of Human Immunodeficiency Virus (HIV) infection or Acquired Immunodeficiency Syndrome (AIDS)-related illness.
2. Active or recent infection (including SARS-COV-2). Participants with prior or recent infection must have infection resolved for >21 days and no use of systemic anti-infective therapy for >28 days.
3. Hepatitis B infection (i.e., hepatitis B surface antigen [HBsAg] or hepatitis B virus [HBV]-DNA positive). In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status.
4. Active hepatitis C infection as measured by positive hepatitis C virus (HCV)-RNA testing. Participants with a history of HCV antibody positivity must undergo HCV-RNA testing. If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCVRNA positive) completed antiviral therapy and has undetectable HCV-RNA for at least 12 weeks following the completion of therapy, the participant is eligible for the study.

   15. Major surgery within 14 days prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment.

NOTE: Participants with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery. If there is a question whether a procedure is considered a major surgery, the Investigator must consult with the appropriate Sponsor representative and resolve any issues before enrolling a participant in the study.

16. Contraindication or intolerance to required supportive care medications in the absence of alternative options.

17. Contraindication or intolerance to daratumumab or lenalidomide, or prior to toxicities to lenalidomide during induction requiring reduction of dose to <10 mg/day.

18. Significant neuropathy (Grades 3-4 or Grade 2 with pain). 19. History of Guillain-Barre Syndrome or variant. 20. Concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures or results, or that in the opinion of the Investigator would constitute a hazard for participating in this study, such as:

1. Uncontrolled diabetes.
2. Acute diffuse infiltrative pulmonary disease.
3. History of autoimmune disease with the exception of vitiligo, type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing.
4. Disabling psychiatric conditions (e.g., alcohol or drug abuse), severe dementia, or altered mental status.
5. Any other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.
6. History of non-compliance with recommended medical treatments.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
Rate of MRD negativity after completion of Maintenance 1 | At 60 weeks
  Rate of participants with MRD negativity (defined as <10-5) after completion of the Maintenance 1 portion of the study.

SECONDARY OUTCOMES:
Rate of sustained MRD negativity after completion of Consolidation and Maintenance 1 or after completion of Maintenance 1 and Maintenance 2 | 60 weeks or 108 weeks, respectively
  Rate of participants with MRD negativity (defined as <10-5) after completion of the Consolidation and Maintenance 1 (negative at both timepoints) or after completion of Maintenance 1 and Maintenance 2 (negative at both timepoints).
Event-free survival (EFS) | 5 years
  Median time from randomization until event using Kaplan-Meier estimates. Event is defined as death, disease progression as defined by the International Myeloma Working Group standard response criteria, initiation of alternative regimen (including Arms A1 or B1 due to MRD positivity after Maintenance 1) or resurgence of MRD (i.e. MRD becoming ≥10-5 after prior negative result <10-5).
Incidence of adverse events | 5 years
  Number of participants with adverse events as assessed by common terminology criteria for adverse events (CTCAE) v5.0.
Rate of MRD negativity at any point in Arm A1 | 72 weeks and 120 weeks, respectively
  Rate of participants with MRD negativity (defined as <10-5) after completion of ASCT or after maintenance treatment.
Rate of MRD negativity at any point in Arm B1 | 72 weeks and 120 weeks, respectively
  Rate of participants with MRD negativity (defined as <10-5) after completion of consolidation with elranatamab and daratumumab or after completion of maintenance with elranatamab and daratumumab.
International Myeloma Working Group (IMWG) Frailty Index- Comparison in participant report outcomes from baseline to end of treatment | 4 years
  Comparison in participant report outcomes from baseline to end of treatment. Frailty score (range 0-5) and categorizes participants into fit (score = 0), intermediate-fit (score = 1) and frail (score ≥ 2).
European Organisation for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire (QLQ)-C30- MY20 module- Comparison in participant report outcomes from baseline to end of treatment | 4 years
  Quality of life questionnaire. Version QLQ-C30. Disease specific module MY-20. Scores are based on a 0-100 scale, with higher scores generally indicating better health-related quality of life.
Patient-Reported Outcomes Measurement Information System (PROMIS)- Comparison in participant report outcomes from baseline to end of treatment | 4 years
  Patient-reported overall health and quality of life questionnaire. Global 10 version. The possible score ranges from 0 to 20 points in each case. 0 points represent the patient's most severe physical and/or mental impairment, while 20 points represent the best possible state of health.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Schade, MD, Study Chair — Colorado Blood Cancer Institute
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Iowa, Iowa City, Iowa
  - University of North Carolina, Chapel Hill, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - Virginia Oncology Associates, Norfolk, Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No